CLINICAL TRIAL: NCT02566850
Title: Investigational Study of the Ekso Bionics Powered Exoskeleton for High-Dosage Use by Individuals With Spinal Cord Injury in a Non-Clinical Environment
Brief Title: Investigational Study of the Ekso for High-Dosage Use by Individuals With SCI in a Non-Clinical Environment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary results acceptable, investigators moved attention to different project
Sponsor: Ekso Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13098
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ekso Users (Experimental): SCI subjects using Ekso
  Interventions: Device: Ekso

INTERVENTIONS:
Device: Ekso — powered lower extremity exoskeleton
  Other Names: Ekso GT

SUMMARY:
The purpose of the study is to study the safety and health effects of using the Ekso Bionics powered exoskeleton device in a home setting over an extended period, ranging from 12-42 months.

DETAILED DESCRIPTION:
This is a 36 month exploratory Investigational Study compliant with the NSF Human Subjects regulations (45 CFR 690) trialing a new device for the SCI populations to aid in ambulatory function in a home setting. Ekso Bionics will enable up to twelve (12) subjects with SCI to use an Ekso device in their home for a 12-month period. Qualified subjects will help Ekso Bionics determine the practical use of the device in the home environment and will enable Ekso Bionics to gather data to develop a device for use in a home environment. The study will require a trained spotter to be present at all times that the device is being used. The study will also evaluate the effectiveness of a non-medically licensed spotter to assist the subject.

ELIGIBILITY:
Inclusion Criteria:

* be an experienced user of the Ekso device with a minimum of 20 hours and no more than 50 hours of device use and require no greater than minimal assist (support of up to 25% body weight) for safe and consistent walking.
* no more than 2 episodes of balance loss per 1 hour training session that require no more than moderate assistance (support of 26% to 50% of body weight)
* participants with more than 50 hours of device experience must agree to a 1 month period of non-use prior to acquisition of baseline measures
* be between 18-65 years of age.
* be able to physically fit into the exoskeleton device.
* be able to tolerate upright standing for up to 60 minutes.
* have sufficient joint range of motion to fit safely within Ekso: Hip flexion contracture ≤ 15o; knee flexion contracture ≤ 10o; ankle dorsiflexion to neutral with no more than 10o of knee flexion.
* have sufficient upper body strength to balance themselves with two arms
* be fluent in English

Exclusion Criteria:

* Height below 60 inches or above 76 inches or with physical characteristics incompatible with device and testing procedure.
* Weight above 220 lbs.
* Lower extremity joint contractures that exceed device capacity for safe use.
* Any medical issue that precludes full weight bearing and ambulation (e.g. osteoporosis that prevents safe standing, orthopedic injuries, pain, severe spasticity)
* Skin integrity issues that would prevent wearing the device.
* Cognitive and/or communicative disability inappropriate for testing as determined by Ekso Bionics clinician. Subjects must be able to follow directions well and demonstrate learning capability.
* Pregnancy (Self-reported)
* Colostomy
* Medical or environmental conditions arising after the start of the study that are deemed unsafe per Ekso Bionics discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ekso Bionics, Richmond, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ekso Users
Started | 4
Completed | 3
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: four males with SCI
Arm/Group | Ekso Users
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39.5 [29 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
ASIA impairment scale (AIS) [Count of Participants; unit: Participants] — A standardized neurological examination to assess the sensory and motor levels which were affected by SCI. Scale has five classification levels, ranging from complete loss of neural function in the affected area to completely normal. Grades are A->E, where E indicates normal and A indicates no sensory or motor function below the level of injury.
  Participants
    AIS A (motor and sensory complete) | 3
    AIS B (motor complete) | 0
    AIS C (incomplete) | 1
    AIS D (incomplete) | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants With Adverse Events
Description: evaluate the safety of a subject walking with a lay spotter in a non-clinical environment
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: International Spinal Cord Injury Data Sets Quality of Life Basic Data Set
Description: Consists of 3 variables: ratings of satisfaction with general quality of life, satisfaction with physical health, and satisfaction with psychological health. All variables are rated on a scale ranging from 0 (completely dissatisfied) to 10 (completely satisfied) with a total of 30 points.
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
score on a scale
  Baseline/Pre intervention | 21 [13 to 30]
  Post intervention up to 42 months | 24.33 [21 to 27]

3. Secondary Outcome: International Spinal Cord Injury Data Sets Bowel Function Basic Data Set
Description: evaluate the impact on subject's bowel health, subjective questionnaire. Examined time required for defecation in minutes, with shorter time being more favorable
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Mean (Full Range); unit: minutes
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
minutes
  time required for defectation - baseline/pre intervention | 28 [6 to 60]
  time required for defectation post intervention up to 42 months | 16.83 [0 to 60]

4. Secondary Outcome: International Spinal Cord Injury Data Sets Bladder Function Basic Data Set - Number of Participants Who Reported Changes in Bladder Function
Description: evaluate the impact on subject's bladder health, subjective feedback and written answers collected, no numerical scoring is part of this exam. This data set asks the following questions: Urinary tract impairment unrelated to spinal cord lesion? Awareness of the need to empty the bladder? How does bladder emptying occur? Average number of voluntary bladder emptyings per 24 hours during the last week? Any involuntary urine leakage (urinary incontinence) within the last four weeks? Collecting appliances for urinary incontinence? Any drugs with possible influence on the urinary tract within the last four weeks? Surgical procedures on the urinary tract? Any change in lower urinary tract symptoms within the last year?
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Spasticity as Tested by the Modified Ashworth Scale
Description: evaluate the impact on subject's spasticity, assessed Elbow Flexors / Extensors, Wrist Flexors / Extensors, Hip Flexors / Extensors, Hip Abductors, Knee Flexors / Extensors, Ankle Plantar Flexors, Ankle Invertors and totaled spasticity for each group (0-5 for right and left) to total between 0 and 70. Higher scores for each muscle group indicate more rigid spasticity, and higher total score indicates more muscle groups involved.
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
units on a scale
  baseline/pre intervention | 0.67 [0 to 2]
  post intervention up to 42 months | 4.67 [0 to 14]

6. Secondary Outcome: International Spinal Cord Injury Data Sets
Description: evaluate the impact on subject's pain. Totaled the following questions with scales from 0-10 for a total score ranging from 0-50. For each question, 0 = "No interference", 10 = "Extreme interference"
  "How much has pain changed your ability to take part in recreational and other social activities?" "How much has pain changed the amount of satisfaction or enjoyment you get from family related activities?" "In general, how much has pain interfered with your day to day activities in the last week?" "In general, how much has pain interfered with your overall mood in the past week?" "In general, how much has pain interfered with your ability to get a good night's sleep?"
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
units on a scale
  baseline/Pre intervention | 13.67 [0 to 27]
  post intervention up to 42 months | 4.67 [0 to 14]

7. Secondary Outcome: Spinal Cord Independence Measure (SCIM) II
Description: evaluate the impact on subject's functional abilities in 3 domains (self care, respiration and sphicter management, mobility) on a scale from 0-100. Each of the 17 total questions have multiple options that are scored in different values. Some questions range from 0-1 points, while others range from 0-2,0-3, 0-5, 0-8, 0-6,0-10, or 0-15. Higher values for each question, and overall, indicate more independence with the task, while lower scores indicates requiring of more assistance.
Time Frame: through study completion for a maximum possible duration of 42 months
Population: One dropout from original 4 participants
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
score on a scale
  baseline/Pre intervention | 71.67 [68 to 75]
  Post intervention up to 42 months | 74 [72 to 76]

8. Secondary Outcome: Strength Via Upper and Lower Extremity Motor Scors (ISNCSCI Exam)
Description: evaluate the impact on subject's muscle strength. Total upper and lower extremity motor scores (0-5 for right and left) for each of the following muscle groups for a total of 120 points. For each muscle group, 0 is defined as no palpable contraction, while 5 is full strength.
  Shoulder Flexion Shoulder Extension Elbow Flexion Elbow Extension Wrist Extension Gross Grip Strength Hip Flexion Hip Extension Hip Abduction Knee Extension Ankle Dorsiflexion Ankle Plantar Flexion
Time Frame: through study completion for a maximum possible duration of 42 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
score on a scale
  baseline/Pre intervention | 69 [60 to 87]
  post intervention up to 42 months | 72.3 [60 to 97]

9. Secondary Outcome: Borg Perceived Rate of Exertion
Description: evaluate the impact on subject's effort while walking. Measure taken for each session on scale from 6-20. Average was taken from each participant over their total number of sessions. Higher scores on the Borg indicates the participants feels like they are working harder.
Time Frame: through study completion for a maximum possible duration of 42 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
score on a scale | 8.98 [7.99 to 10.93]

10. Secondary Outcome: Length of Participation in Study
Description: Number of months that a participant utilized the Ekso in their home with a lay spotter
Time Frame: through study completion for a maximum possible duration of 42 months
Population: one dropout
Measure: Mean (Full Range); unit: months
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
months | 31.67 [15 to 42]

11. Secondary Outcome: Secondary Health Conditions
Description: Frequency of secondary health complications as reported by participants
Time Frame: Through study completion for a maximum possible duration of 42 months
Population: one dropout
Measure: Count of Participants; unit: Participants
Arm/Group | Ekso Users
Number analyzed (Participants) | 3
Participants
  Participants who reported a UTI during study duration | 0
  Participants who reported a pressure sore during study duration | 0
  Participants who reported no secondary health conditions during study duration | 3

ADVERSE EVENTS:
Time Frame: Through completion of the study, which could be up to 42 months
Arm/Group | Ekso Users
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT02566850/Prot_000.pdf
  • Informed Consent Form (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT02566850/ICF_001.pdf